CLINICAL TRIAL: NCT07025304
Title: A Prospective, Multi-center, Post-Market Clinical Study to Evaluate the Safety and Effectiveness of the REFLEX ULTRA 45 for the Coblation Inferior Turbinate Reduction in China
Brief Title: Post-Market Clinical Study to Evaluate the Safety and Effectiveness of REFLEX ULTRA 45 for Coblation Inferior Turbinate Reduction in China
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Smith & Nephew, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SNIS-E-1198
Record Dates: First submitted 2025-06-09; First posted 2025-06-17 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2025-07

CONDITIONS: Nasal Obstruction Due to Inferior Turbinate Hypertrophy
Keywords: REFLEX; CITR; ITH; Coblation Inferior Turbinate Reduction; Inferior Turbinate Hypertrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- REFLEX ULTRA 45 (Experimental): The investigational product REFLEX ULTRA 45 includes two models which are EIC4845-01 and EICA4845-01. The only difference between these two models is the EICA4845-01 has a maximum two-use limit.
  Interventions: Device: REFLEX ULTRA 45

INTERVENTIONS:
Device: REFLEX ULTRA 45 — One time use for surgery

SUMMARY:
The study is a prospective, multi-center, post-market clinical study to evaluate the safety and effectiveness of REFLEX ULTRA 45 for the coblation inferior turbinate reduction in China. The study product is REFLEX ULTRA 45 (EIC4845-01/EICA4845-01). Also it needs to be performed with the controller system COBLATOR II or WEREWOLF. The sample size is 105 subjects with approximate 6 sites in China mainland.

DETAILED DESCRIPTION:
Inferior turbinate hypertrophy (ITH) is a common condition characterized by the enlargement of the inferior turbinate which is mainly due to swelling of the sub-mucosa and rarely due to enlargement of the bone itself. Based on current studies, there are several surgical techniques is being widely used in clinic for ITH includes turbinectomy, electrocautery, laser surgery, cryotherapy, Microdebrider-assisted inferior turbinoplasty (MAIT) and radiofrequency ablation (RFA). The technique used in this study for ITH is Coblation produced by REFLEX ULTRA 45. With limited high quality literature in Chinese population, it is the main purpose to generate high quality evidence among the Chinese population to establish the effectiveness and safety in Chinese population with sufficient outcomes evaluation and appropriate inclusion and exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Subject with at least two-year history of perennial rhinitis and who has failed one month of continuous standardized treatment with hormonal nasal spray by the date of surgery.
* Subject with nasal obstruction due to turbinate hypertrophy and is suitable to receive coblation inferior turbinate reduction for bilateral nasal cavity without outfracture of inferior turbinate per the investigator's judgement.
* Subject is 18 - 65 years old (inclusive).
* Subject provides written informed consent for study participation using an Independent Ethical Committee (IEC) approved consent form before any study procedures are performed, including pre- operative data review and/or collection of data on electronic Case Report Forms (eCRFs).
* Subject is willing and able to participate in required follow-up visits and is able to complete study activities.

Exclusion Criteria:

* Subject who does not meet the indication or is contraindicated according to specific REFLEX ULTRA 45 's Instructions for Use (IFUs).
* Subject with obvious deviation of nasal septum with the necessity of surgery under investigator's judgement.
* Participation in the treatment period of another clinical trial within thirty (30) days of all visits completed.
* Subject who needs other nasal surgery other than single inferior turbinate reduction evaluated by MRI and nasal endoscopy.
* Subject who has nasal obstruction due to inferior turbinate bony hypertrophy.
* Subject who was treated with inferior turbinate reduction before informed consent.
* Subjects who completed the Zung Self-Rating Anxiety Scale and the anxiety rate is more than 59.
* Woman who is pregnant, nursing, or of child-bearing potential who are not utilizing highly effective birth control measures.
* Any subject that meets the definition of a Vulnerable Subject per ISO 14155 Section 3.55.
* Subject who has participated previously in this clinical trial or who has been withdrawn.
* Subject with a history of poor compliance with medical treatment.
* Subject with a medical or physical condition that, in the opinion of the Investigator, would preclude safe subject participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2025-07-02 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Nasal Obstruction Symptom Evaluation (NOSE) score at 3 Months | 3 months
  Nasal Obstruction Symptom Evaluation (NOSE) consists of 5 questions regarding nasal congestion or stuffiness, nasal blockage or obstruction, trouble breathing through nose, trouble sleeping, and ability to get enough air through nose during exercise or exertion. NOSE scores range from 0 to 100, with a higher score indicating a severe problem (i.e., worse outcome) and lower score indicating no problem (i.e., better outcome).

SECONDARY OUTCOMES:
Nasal Obstruction Symptom Evaluation (NOSE) score | 7 days, 1 month, 6 months, 1 year, 2 years
  Nasal Obstruction Symptom Evaluation (NOSE) consists of 5 questions regarding nasal congestion or stuffiness, nasal blockage or obstruction, trouble breathing through nose, trouble sleeping, and ability to get enough air through nose during exercise or exertion. NOSE scores range from 0 to 100, with a higher score indicating a severe problem (i.e., worse outcome) and lower score indicating no problem (i.e., better outcome).
36-Item Short Form Survey (SF-36) | 7 days, 3 months, 1 year, 2 years
  The 36-Item short form survey instrument taps eight health concepts: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. It also includes a single item that provides an indication of perceived change in health. Possible scores range from 0 to 100 for each item, with higher scores indicating a better outcome.
Unilateral Nasal Resistance | 3 months, 1 year, 2 years
  Nasal resistance is an objective indicator of nasal respiratory function, measured using a rhinomanometry device. During the assessment, the participant breathes air into a tube connected to the rhinomanometry device. The device measures the air pressure and rate of airflow, which are then used to calculate nasal resistance. Increased nasal resistance values indicate nasal obstruction. Unilateral nasal resistance measures the resistance to airflow through one nostril at a time.
Total Nasal Resistance | 3 months, 1 year, 2 years
  Nasal resistance is an objective indicator of nasal respiratory function, measured using a rhinomanometry device. During the assessment, the participant breathes air into a tube connected to the rhinomanometry device. The device measures the air pressure and rate of airflow, which are then used to calculate nasal resistance. Increased nasal resistance values indicate nasal obstruction. Total nasal resistance measures the combined resistance to airflow through both nostrils simultaneously.
Minimal Cross-Sectional Area | 3 months, 1 year, 2 years
  Minimal cross-sectional area (MCA) of the nasal passage will be measured using acoustic rhinometry. This technique provides detailed information on the geometry of the nasal cavity, identifying the narrowest part of the airway. MCA values will be recorded in square centimeters (cm^2) to assess how open the nasal passages are and potential obstructions.
Nasal Volume | 3 months, 1 year, 2 years
  Nasal volume of the nasal cavity will be measured using acoustic rhinometry. Acoustic rhinometry is a standard diagnostic tool in objective evaluation of nasal patency. The information on the geometry of nasal cavities is provided using acoustic waves generated by the acoustic rhinometry device. It is an easy and non-painful procedure to perform. By placing a nosepiece into patient's nostril and performing breath holding, the information on the structure and dimensions of the nasal cavity is captured. Nasal volume values will be recorded in cubic centimeters (cm^3) to assess how open the nasal cavity is and potential obstructions.
Mucociliary Transport Function Time | 3 months, 1 year, 2 years
  Mucociliary transportation function will be measured using a saccharin test. During this test a saccharin particle measuring 1mm in diameter is placed under direct vision, on the medial surface of the interior nasal turbinate. The time taken for the participant's initial perception of the sweet taste of saccharin will be recorded in minutes.
Mucociliary Transport Function Distance | 3 months, 1 year, 2 years
  Mucociliary transportation function will be measured using a saccharin test or endoscopy. The distance from the saccharin placement site to the posterior wall of the pharynx could be measured by inserting a long cotton swab into the posterior wall of the nasopharynx of subject or nasal endoscopy.
Surgeon Evaluation of Turbinate/Mucosal Tissue Health - Inferior Turbinate Hypertrophy Grade by Anterior Rhinoscopy | 7 days
  Anterior rhinoscopy is performed as a part of physical examination of turbinate/mucosal tissue health. The doctor wears a headlight to free up the hands and shines the light into the nose. A speculum is introduced into the nasal vestibule by the doctor to observe inferior turbinate, inferior meatus, and the upper part of the nasal cavity.
  The anterior rhinoscopic assessment will help evaluate nasal mucosa, sinonasal anatomy and nasal pathology. Inferior turbinate hypertrophy assessed by anterior rhinoscopy to identify the degree of nasal obstruction will be categorized as one of the following grades:
  * Grade 1: The inferior turbinate occupied less than half of the nasal cavity and no obvious nasal obstruction was observed
  * Grade 2: Hypertrophied inferior turbinate occupied more than 50% of the nasal cavity
  * Grade 3: A complete occlusion of the nasal cavity occurred because of the severe enlargement of the inferior turbinate
Surgeon Evaluation of Turbinate/Mucosal Tissue Health - Presence of Crusting and Bleeding by Anterior Rhinoscopy | 7 days
  Anterior rhinoscopy is performed as a part of physical examination of turbinate/mucosal tissue health. The doctor wears a headlight to free up the hands and shines the light into the nose. A speculum is introduced into the nasal vestibule by the doctor to observe inferior turbinate, inferior meatus, and the upper part of the nasal cavity.
  The anterior rhinoscopic assessment will help evaluate nasal mucosa, sinonasal anatomy and nasal pathology. Anterior rhinoscopy will be used to identify the presence of crusting and bleeding (Yes/No).
Surgeon Evaluation of Turbinate/Mucosal Tissue Health - Inferior Turbinate Hypertrophy Grade by Nasal Endoscopic Assessment | 3 months, 1 year, 2 years
  Endoscope is a thin, flexible, or rigid tube with a tiny camera and a light. During the procedure, the doctor will put the endoscope into the patient's nose and guide it through the nasal and sinus passages. Image of the area is seen through the endoscope which helps evaluate nasal mucosa, sinonasal anatomy and nasal pathology.
  Inferior turbinate hypertrophy assessed by the nasal endoscopic assessment to identify the degree of nasal obstruction will be categorized as one of the following grades:
  * Grade 1: The inferior turbinate occupied less than half of the nasal cavity and no obvious nasal obstruction was observed
  * Grade 2: Hypertrophied inferior turbinate occupied more than 50% of the nasal cavity
  * Grade 3: A complete occlusion of the nasal cavity occurred because of the severe enlargement of the inferior turbinate
Surgeon Evaluation of Turbinate/Mucosal Tissue Health - Magnetic Resonance Imaging (MRI) | 3 months, 1 year, 2 years
  MRI on the nasal cavity or paranasal sinuses will be used to evaluate turbinate/mucosal tissue health to identify presence of sinusitis, tumors, polyps, and deformities.
Duration of Surgery | During procedure
  The time of surgery from start to end will be recorded.
Intraoperative Bleeding | During procedure
  The blood loss during surgery will be categorized as one of the following: 0-5ml, 5-15ml or>15ml

CONTACTS AND LOCATIONS:
Overall Officials: Dongdong Zhu, Principal Investigator — China-Japan Union Hospital, Jilin University
Locations (6):
- China (6):
  - The First Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - The Third Affiliated Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - China-Japan Union Hospital of Jilin University, Changchun, Jilin
  - Sir Run Run Shaw Hospital Affiliated with Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No